CLINICAL TRIAL: NCT03506308
Title: A Prospective, Global, Multicenter, Single Arm Post-Approval Study Investigating the Clinical Use and Safety of the Lutonix® Drug Coated Balloon PTA Catheter for the Treatment of Dysfunctional AV Fistulae
Brief Title: Post Approval Study Investigating Lutonix Drug Coated Balloon for Treatment of Dysfunctional Arteriovenous Fistulae
Acronym: AVPAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL0033-01
Record Dates: First submitted 2018-04-14; First posted 2018-04-24 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- LUTONIX 035 Drug Coated Balloon PTA Catheter (Other): This is a single-arm study. All subjects will receive the Lutonix® 035 Drug Coated Balloon PTA Catheter.
  Interventions: Device: LUTONIX 035 Drug Coated Balloon PTA Catheter

INTERVENTIONS:
Device: LUTONIX 035 Drug Coated Balloon PTA Catheter — All subjects will receive the Lutonix® 035 Drug Coated Balloon PTA Catheter.

SUMMARY:
This prospective, global, multicenter, single arm post-approval study is designed to investigate the clinical use and safety of the Lutonix® 035 AV Drug Coated Balloon (DCB) PTA Catheter in subjects presenting with clinical and hemodynamic abnormalities in native arteriovenous (AV) fistulae located in the upper extremity.

DETAILED DESCRIPTION:
This post-market approval study (PAS) is required by the FDA as a condition of approval for the Lutonix drug coated balloon catheter. It is intended to demonstrate safety and assess the clinical use and outcomes of the LUTONIX Catheter in dysfunctional arteriovenous fistulae (AVF) in a heterogeneous patient population in real world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-breastfeeding female ≥18 years of age
2. Subject is willing to provide informed consent, and is willing to comply with the protocol-required follow up visits
3. Target lesion must be a mature arteriovenous fistula located in the arm presenting with any clinical, physiological or hemodynamic abnormalities warranting angiographic imaging as defined in the K/DOQI guidelines
4. Subject has a target lesion that can be treated with available LUTONIX DCB according to the Instructions For Use (IFU)
5. Venous stenosis of an AV fistula in which the target lesion is located from the anastomosis to the axillosubclavian junction, as defined by insertion of the cephalic vein
6. Successful pre-dilation of the target lesion with an uncoated percutaneous transluminal angioplasty (PTA) balloon defined as:

   1. No clinically significant dissection;
   2. No extravasation requiring treatment;
   3. Residual stenosis ≤30% by angiographic measurement;
   4. Ability to completely efface the waist using the pre-dilation balloon.

Exclusion Criteria:

1. Subject is currently participating in an investigational drug, biologic, or device study, or previous enrollment in this study
2. Subject has a non-controllable allergy to contrast
3. Subject has another medical condition that, in the opinion of the Investigator, may confound the data interpretation or is associated with a life expectancy insufficient to allow for completion of subject study procedure and follow up
4. Target lesion is located central to the axillosubclavian junction
5. A thrombosed access or an access with a thrombosis treated ≤7 days before to the index procedure
6. Prior surgical interventions of the access site ≤30 days before the index procedure
7. Target lesion is located within a bare metal or covered stent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Target Lesion Primary Patency (TLPP) | 6 Months
  TLPP is defined as the interval following index procedure intervention until clinically driven reintervention of the target lesion or access thrombosis.
Percentage of Participants With No Primary Safety Events | 30 days
  Primary safety events include any serious adverse event(s) involving the AV access circuit through 30 days

SECONDARY OUTCOMES:
Percentage of Participants With Target Lesion Primary Patency | 12, 18, 24 Months
  TLPP is defined as the interval following index procedure intervention until clinically driven reintervention of the target lesion or access thrombosis.
Number of re-interventions required to maintain target lesion patency | 6, 12, 18, 24 Months
  Clinically driven reintervention is defined as a lesion that has ≥ 50% stenosis and at least one clinical, physiological or hemodynamic abnormality attributable to the stenosis defined in the K/DOQI guidelines.
Percentage of Participants With Access Circuit Primary Patency (ACPP) | 6, 12, 18, 24 Months
  Access circuit is defined as the area from the AV access anastomosis to the superior vena cava-right atrial junction.
Number of re-interventions required to maintain access circuit patency | 6, 12, 18, 24 Months
  Clinically driven reintervention is defined as a lesion that has ≥ 50% stenosis and at least one clinical, physiological or hemodynamic abnormality attributable to the stenosis defined in the K/DOQI guidelines.
Percentage of Participants With Device, Procedural, and Clinical Success | 24 Months
  Device Success: Successful delivery to the target lesion, deployment, and retrieval at index procedure.
  Procedural Success: At least one indicator of hemodynamic success (e.g., physical examination with restoration of a thrill, direct measurement of flow) in the absence of peri-procedural (index procedure and through hospital stay) Serious Adverse Device Effects (SADEs).
  Clinical Success: The resumption of dialysis for at least one session after the index procedure.
Percentage of Participants With Abandonment of Permanent Access in the Index Extremity | 6, 12, 18, 24 Months
  The arteriovenous fistula / access circuit is considered abandoned when it is no longer being used for dialysis because the access was not functioning.
Percentage of Participants With Secondary Patency of the Access Circuit | 6, 12, 18, 24 Months
  Survival of patency of access circuit from the time of intervention until access abandonment or achievement of a censored event (death, transfer to another hemodialysis unit, transfer to peritoneal dialysis, transplantation, and end of study period), and includes all surgical and endovascular interventions.
Time to loss of target lesion secondary patency following DCB intervention | 24 Months
  Time between first reintervention with the DCB to the next loss of patency
Percentage of Participants With Freedom from any Serious Adverse Event(s) Involving the AV Access Circuit | 6, 12, 18, 24 Months
  Safety events include any serious adverse event(s) involving the AV access circuit
Percentage of Participants With Device and Procedure Related Adverse Events | 6, 12, 18, 24 Months
  Freedom from device-related or procedure-related serious adverse events

OTHER OUTCOMES:
Vital status of participants | 36, 48, and 60 Months
  All cause death

CONTACTS AND LOCATIONS:
Overall Officials: Scott Trerotola, MD, Principal Investigator — Hospital of the University of Pennsylvania; Division of Interventional Radiology; Dheeraj Rajan, MD, Principal Investigator — University Health Network; Division of Vascular & Interventional Radiology
Locations (26):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Flowers Hospital, Dothan, Alabama
  - St. Joseph Hospital of Orange, Orange, California
  - Kaiser Permanente, San Diego, California
  - Yale University, New Haven, Connecticut
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Ochsner Health System, New Orleans, Louisiana
  - Ochsner Louisiana State University Health, Shreveport, Louisiana
  - MedStar Health Research Institute, Annapolis, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Dallas Vascular Center, Dallas, Texas
  - HCA Houston Healthcare, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center, Houston, Texas
  - Sentara Medical Group, Norfolk, Virginia
- Canada (4):
  - William Osler Health System/Brampton Civic Hospital, Brampton, Ontario
  - Scarborough Health Network, Scarborough Village, Ontario
  - University Health Network, Toronto, Ontario
  - Centre hospitalier de l'Université de Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No